

UCLH Project ID number: 07/Q0502/15 Form version 5, 7<sup>th</sup> February 2023

## **Imaging Department**

University College London Hospital 235 Euston Road London NW1 2BU

Telephone: 020 3456 7890 ext 73283

Website: www.uclh.nhs.uk

UCLH Project ID number: 07/Q0502/15 Form version 5, 7<sup>th</sup> February 2023

## **CONSENT FORM**

Title of project: Development of novel magnetic resonance techniques using volunteer participants.

Name of Principal Investigator: Professor Shonit Punwani

| 1. | I confirm that I have read and understood the patient information sheet dated 7 <sup>th</sup> February 2023 (version 7) for the above study and have had the opportunity to ask questions. | Please initial each box |
|---|---|---|
| 2. | I confirm that I have had sufficient time to consider whether or not want to be included in the study. | |
| 3. | I understand that my participation is voluntary and that I am free to withdraw at any time, without giving any reason, without my medical care or legal rights being affected. | |
| 4. | I agree to the administration of a contrast agent for this research. | |
| 5. | I understand that this research scan is not intended for diagnostic purposes. In the unlikely event that something on the scan suggests a need for medical follow-up, I understand that a radiologist will inform me, and may contact my GP if appropriate. | |
| 6. | I agree to allow any MRI data acquired during my scan to be used, anonymised so that I cannot be identified, for research or teaching. | |
| 7. | I agree to take part in the above study. | |
| (C | ontinued overleaf) | |

UCL Hospitals is an NHS Trust incorporating the Elizabeth Garrett Anderson & Obstetric Hospital, Hospital for Tropical Diseases, Institute of Sport, Exercise and Health, National Hospital for Neurology & Neurosurgery, The Royal London Hospital for Integrated Medicine, Royal National ENT and Eastman Dental Hospitals, University College Hospital, University College Hospital at Westmoreland Street, University College Hospital Grafton Way Building and University College Hospital Macmillan Cancer Centre.



UCLH Project ID number: 07/Q0502/15 Form version: 5, 7<sup>th</sup> February 2023

## **CONSENT FORM**

Title of project: Development of novel magnetic resonance techniques using volunteer participants.

Name of Principal Investigator: Professor Shonit Punwani

This study has no diagnostic purpose and is not intended for screening or diagnostic purposes. However, in the unlikely event that something on the scans suggests a need for medical follow-up, a radiologist will review the images and inform you. They may also contact your GP.

| Name of volunteer | Date | Signature |
|---|---|---|
| Name of person taking consent | <br>Date | Signature |
| Researcher to contact if there are a | any problems (nam | ne, organisation and telephone |
| number): | | |

## Comments or concerns during the study

If you have any comments or concerns you may discuss these with the investigator. If you wish to go further and complain about any aspect of the way you have been approached or treated during the course of the study, you should contact the UCLH Patient Advice and Liaison Service (PALS) the details of whom are on the patient information sheet. Please quote the UCLH project number at the top this consent form.